CLINICAL TRIAL: NCT04761770
Title: Phase II Study of a Geriatric Assessment-Driven, Risk-Adapted Allogeneic Hematopoietic Cell Transplant Strategy for Older Patients With Myeloid Malignancies
Brief Title: Study of a Geriatric Assessment to Plan a Treatment Approach for Older People With Various Blood Disorders
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-522
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Myelodysplastic Syndrome; Myeloproliferative Neoplasms; Chronic Myelomonocytic Leukemia; Atypical Chronic Myeloid Leukemia; Myelodysplastic/Myeloproliferative Overlapping Syndrome
Keywords: blood disorders; Allogeneic Hematopoietic Cell Transplant; 20-522
MeSH Terms: conditions — Myelodysplastic Syndromes; Myeloproliferative Disorders; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Hematologic Diseases | interventions — Geriatric Assessment; Transplantation Conditioning

STUDY DESIGN:
Intervention Model Description: This is a prospective, single center, phase II pilot treatment-allocation study at MSK for older patients considering allogeneic hematopoietic cell transplantation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Geriatric participants with various blood disorders (Experimental): 1. Geriatric assessment (GA) pre-transplant
  2. Risk-adapted allocation of conditioning intensity based on GA
  3. GA-directed, longitudinal supportive care management
  Interventions: Other: Geriatric assessment (GA) pre-transplant; Drug: conditioning regimen; Procedure: Allogeneic CD34+ selected stem cells

INTERVENTIONS:
Other: Geriatric assessment (GA) pre-transplant — Assessment of comorbidities, polypharmacy, and functional, nutritional, and psychosocial impairment.
Drug: conditioning regimen — Based on the Geriatric assessment.
  1. HCT-CI/Age ≤4 AND no IADL impairment (less vulnerable/fit) -> Myeloablative (MA) regimen
  2. HCT-CI/Age >4 AND/OR any IADL impairment (more vulnerable) -> Reduced-intensity (RIC)/Nonmyeloablative (NMA) regimen
Procedure: Allogeneic CD34+ selected stem cells — Stem cells are collected as per institutional guidelines. CD34+ enriched stem cells will be obtained using the FDA approved reagents from Miltenyi, according to the instruction manual.

SUMMARY:
This study will evaluate whether a geriatric assessment can lead to better treatment outcomes in older patients (age 60+) with a myeloid malignancy including acute myeloid leukemia, ,myelodysplastic syndromes, myeloproliferative neoplasms, or related blood disorders who are going to receive chemotherapy or another treatment to prepare the body for an allogeneic hematopoietic stem cell transplant (allo-HCT). The geriatric assessment includes looking at patients' cognitive function (thinking processes), physical function, mobility (ability to move the body), mood, nutrition, and current medications to help decide the type of treatment they'll receive.

Another purpose of this study is to see whether use of the geriatric assessment improves participants' quality of life. We will evaluate participants' quality of life through questionnaires.

DETAILED DESCRIPTION:
This is a prospective, phase II study evaluating the efficacy of a risk-adapted, personalized allo-HCT strategy based on geriatric vulnerabilities identified by pre-transplant GA. The less vulnerable/fit older patients are recommended to receive MA conditioning and the more vulnerable older patients are recommended to receive RIC/NMA conditioning.

1. HCT-CI/Age ≤4 AND no IADL impairment (less vulnerable/fit) -> MA regimen
2. HCT-CI/Age >4 AND/OR any IADL impairment (more vulnerable) -> RIC/NMA regimen

   * Chemotherapies: busulfan, fludarabine, melphalan, cyclophosphamide, thiotepa, clofarabine
   * Radiation therapy: total body irradiation (TBI)
   * Other therapy: anti-thymocyte globulin (ATG)

ELIGIBILITY:
Inclusion Criteria:

* are 60 years or older
* have a pathologically confirmed myeloid malignancies including acute myeloid leukemia, ,myelodysplastic syndrome, myeloproliferative neoplasms, or related blood disorders including chronic myelomonocytic leukemia, atypical chronic myeloid leukemia, and myelodysplastic/myeloproliferative overlapping syndrome
* have <10% blasts in bone marrow prior to transplant
* have a matched related or unrelated donor, mismatched unrelated donor, or haploidentical donor
* Meet institutional standard criteria for allogeneic transplantation as determined by the primary transplant physician
* Undergoes transplantation using the allocated conditioning regimen intensity defined by the protocol-specified criteria below:

  * HCT-CI/Age <5 and IADL normal = myeloablative regimen
  * HCT-CI/Age ≥5 and/or IADL impairment = RIC/NMA regimen

Exclusion Criteria:

* Prior hematopoietic cell transplantation
* Cord blood donors
* Persons with active, refractory disease defined by ≥10% blasts in bone marrow prior to transplant

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
cumulative incidence of non-relapse mortality (NRM) | 1 year
  defined as death in the absence of relapse/disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Lin, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent Only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent Only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Consent Only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm